CLINICAL TRIAL: NCT03143803
Title: Control of Glycemic Variability Using a Polyherbal: A Randomized Placebo Controlled Study of Whole Herb Formulations
Brief Title: Control of Blood Glucose Fluctuation With Usage of Polyherbal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OI-005-2017
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyherbal (Active Comparator): Polyherbal capsule contains leaves of 3 herbs namely C. indica, B. spectabilis and C. rosea.
  Interventions: Drug: Polyherbal capsule coccinia, bougainvillea, catharanthus
- Placebo (Placebo Comparator): Placebo will contain an inert substance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyherbal capsule coccinia, bougainvillea, catharanthus — A unique combination of 3 herbs that lower blood sugars
  Other Names: Sugar Balance (SB)
  Arms: Polyherbal
Drug: Placebo — Similar looking inactive powder
  Arms: Placebo

SUMMARY:
The aim of the study is to get insight into control of glycemic variability with Sugar Balance capsules which is the leaves of three herbs: ivy ground (Coccinia indica)-200mg, bougainvillia (Bougainvillea spectabilis)-30mg, Madagascar periwinkle (Catharanthus rosea)-20mg.

DETAILED DESCRIPTION:
The glycemic variability would be obtained at 14 days with the usage of Flash glucose monitoring system manufactured by Abbott and outcomes would be compared at the end of ambulatory glucose profile.

ELIGIBILITY:
Inclusion Criteria:

Adult males and non-pregnant females aged ≥18 years having a diagnosis of pre-diabetes (impaired fasting glucose or impaired glucose tolerance) or diabetes and meeting one of the following criteria

1. Fasting Plasma Glucose ≥100 mg/dL, fasting defined as no caloric intake for at least 8 hours, AND
2. Glycosylated haemoglobin (A1C) ≥ 6 %. The test should be performed in a laboratory using a method that is National Accreditation Board for Testing and Calibration Laboratories certified and standardized within last 3 months.

Exclusion Criteria:

Any one of the following

1. Patients on Insulin therapy.
2. Any history suggestive of micro vascular or macro vascular disease - coronary artery disease, stroke, peripheral artery disease or diabetes related retinal changes.
3. Women in child bearing age unable to practice any form of contraception
4. Patients with diagnosis of Anemia (Hb<11 g/dl in Female and <13 g/dl in Male)
5. Impaired renal function; estimated estimated glomerular filtration rate <60mls/min/1.73m2.
6. Known history of any chronic illness taking regular pharmacological agents.
7. Blood pressure fluctuations exceeding 20 mm of Hg on 2 subsequent clinic visits or known history of hypo tension or bradycardia in last 6 months or taking 3 or more anti-hypertensive medications regularly in the last 6 weeks
8. Known history of autonomic dysfunction like diabetic autonomic neural imbalance or neuropathy
9. Current or former employees of organic India or any potential conflict of interest in participation
10. Participating in another clinical trial with an active intervention or drug or device with last dose taken within 60 days.
11. Refusing consent or physician uncomfortable with patient compliance to treatments or follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Mean amplitude glycemic excursion | 14 days
  To demonstrate that the difference in mean amplitude glycemic excursions among patients receiving polyherbal medication will be less than 1mmol/dL or 18mg/dL for a sampling frequency: 1 every 15 minutes over 14 days

SECONDARY OUTCOMES:
Mean estimated glycated hemoglobin | 14 days
  Mean estimated glycated hemoglobin difference between test and placebo control group
Number of hypoglycemia episodes | 14 days
  Number of hypoglycemia episodes and duration of hypoglycemia in treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Alben Sigamani, Principal Investigator — Narayana Hrudayalaya Hospital
Locations (1):
- Mazumdar Shaw Medical Centre, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided